CLINICAL TRIAL: NCT01059071
Title: A Phase I Trial for Refractory or Relapsed Neuroblastoma With DFMO Alone and in Combination With Etoposide
Brief Title: Safety Study for Refractory or Relapsed Neuroblastoma With DFMO Alone and in Combination With Etoposide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Giselle Sholler (Other)
Collaborators: Cancer Prevention Pharmaceuticals, Inc. (Industry); University of Arizona (Other); University of Hawaii (Other)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMTRC 002
Record Dates: First submitted 2010-01-26; First posted 2010-01-29 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Neuroblastoma
Keywords: Refractory Neuroblastoma; Relapsed neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Eflornithine; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DFMO and Etoposide (Experimental)
  Interventions: Drug: DFMO; Drug: Etoposide

INTERVENTIONS:
Drug: DFMO — Escalating doses of DFMO in a 3 +3 cohort design.
  DFMO at current cohort Dose Level orally each day for 21 day cycles
  Dose level 1: 500 mg/m2 PO BID Dose level 2: 750 mg/m2 PO BID Dose level 3:1000 mg/m2 PO BID Dose level 4:1500 mg/m2 PO BID
  Other Names: Difluoromethylornithine
Drug: Etoposide — Starting with Cycle 2, etoposide will be given at 50mg/m2/dose PO daily for the first 14 days of each 21 day cycle. Capsules will be rounded to closest 50 mg.
  Other Names: Eposin; Etopophos; Vepesid; VP-16

SUMMARY:
The purpose of this research study is to evaluate a new investigational drug to treat neuroblastoma. This study drug is called DFMO. The objectives of this study will be to monitor for safety and to find a maximum tolerated dose in this population. A secondary objective will be to look at efficacy of DFMO.

The safety of the proposed dosing regimen in this trial will be tested by an on-going risk/benefit assessment during the study. A patient benefiting from treatment, not progressing on therapy, and in the absence of any safety issues associated with DFMO and/or etoposide may continue on treatment with the expectation that there will be an overall clinical benefit.

The procedures involved in this study include Medical history, Physical exam, Vital signs (blood pressure, pulse, temperature), Blood tests, Urine tests, MRI or CT scan of the tumor(s), MIBG scans, and Bone marrow aspirations. All of these tests and procedures are considered standard of care for this population. Drug administration is also part of this protocol, including an investigational new drug called DFMO, and later combined with an already approved drug, etoposide.

The proposed dosing regimen is an oral dose of DFMO two times a day for each day while on study. There will be 5 cycles. Each cycle will be 21 days in length. The first cycle will be DFMO alone. In the second cycle etoposide will be added in and will be given orally once a day for the first 14 days of each cycle (cycles 2-5).

ELIGIBILITY:
Inclusion Criteria:

* Age: 0-21 years at the time of diagnosis.
* Diagnosis: Histologic verification at either the time of original diagnosis or relapse of neuroblastoma.
* Disease Status: Refractory or relapsed neuroblastoma
* Measurable disease, including at least one of the following:

Measurable tumor >10mm by CT or MRI A positive MIBG and abnormal urinary catecholamine levels Positive bone marrow biopsy/aspirate.

* Current disease state must be one for which there is currently no known curative therapy.
* A negative urine pregnancy test is required for female subjects of child bearing potential (onset of menses or ≥13 years of age).
* Patients without bone marrow metastases must have an ANC > 500/μl and platelet count >50,000/μl
* Organ Function Requirements Subjects must have adequate liver function as defined by AST or ALT <10x normal Serum bilirubin must be ≤ 2.0 mg/dl Serum creatinine must be ≥ 1.5 mg/dl
* Informed Consent: All subjects and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Life expectancy <2 months or Lansky score <30%
* Investigational Drugs: Subjects who are currently receiving another investigational drug are excluded from participation.
* Anti-cancer Agents: Subjects who are currently receiving other anticancer agents are not eligible. Subjects must have fully recovered from the effects of prior chemotherapy (hematological and bone marrow suppression effects)
* Infection: Subjects who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
* Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-02; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer at Atrium Health
Locations (7):
- United States (7):
  - Children's Hospital of Orange County, Orange, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Arnold Palmer Hospital for Children- MD Anderson, Orlando, Florida
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Levine Children's Hospital, Charlotte, North Carolina
  - UVM/FAHC, Burlington, Vermont

REFERENCES:
- [Derived] Saulnier Sholler GL, Gerner EW, Bergendahl G, MacArthur RB, VanderWerff A, Ashikaga T, Bond JP, Ferguson W, Roberts W, Wada RK, Eslin D, Kraveka JM, Kaplan J, Mitchell D, Parikh NS, Neville K, Sender L, Higgins T, Kawakita M, Hiramatsu K, Moriya SS, Bachmann AS. A Phase I Trial of DFMO Targeting Polyamine Addiction in Patients with Relapsed/Refractory Neuroblastoma. PLoS One. 2015 May 27;10(5):e0127246. doi: 10.1371/journal.pone.0127246. eCollection 2015. PMID 26018967
- See also: Beat Childhood Cancer Consortium website — http://www.beatcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 500 mg/m2 PO BID: DFMO: Escalating doses of DFMO in a 3 +3 cohort design.
  DFMO at current cohort Dose Level orally each day for 21 day cycles
  Dose level 1: 500 mg/m2 PO BID
  Etoposide: Starting with Cycle 2, etoposide will be given at 50mg/m2/dose PO daily for the first 14 days of each 21 day cycle. Capsules will be rounded to closest 50 mg.
- Dose Level 2: 750 mg/m2 PO BID: DFMO: Escalating doses of DFMO in a 3 +3 cohort design.
  DFMO at current cohort Dose Level orally each day for 21 day cycles
  Dose level 2: 750 mg/m2 PO BID
  Etoposide: Starting with Cycle 2, etoposide will be given at 50mg/m2/dose PO daily for the first 14 days of each 21 day cycle. Capsules will be rounded to closest 50 mg.
- Dose Level 3:1000 mg/m2 PO BID: DFMO: Escalating doses of DFMO in a 3 +3 cohort design.
  DFMO at current cohort Dose Level orally each day for 21 day cycles
  Dose level 3:1000 mg/m2 PO BID
  Etoposide: Starting with Cycle 2, etoposide will be given at 50mg/m2/dose PO daily for the first 14 days of each 21 day cycle. Capsules will be rounded to closest 50 mg.
- Dose Level 4:1500 mg/m2 PO BID: DFMO: Escalating doses of DFMO in a 3 +3 cohort design.
  DFMO at current cohort Dose Level orally each day for 21 day cycles
  Dose level 4:1500 mg/m2 PO BID
  Etoposide: Starting with Cycle 2, etoposide will be given at 50mg/m2/dose PO daily for the first 14 days of each 21 day cycle. Capsules will be rounded to closest 50 mg.
Period: Overall Study
Arm/Group | Dose Level 1: 500 mg/m2 PO BID | Dose Level 2: 750 mg/m2 PO BID | Dose Level 3:1000 mg/m2 PO BID | Dose Level 4:1500 mg/m2 PO BID
Started | 4 | 5 | 3 | 9
Completed | 2 | 1 | 1 | 3
Not Completed | 2 | 4 | 2 | 6
Not completed — Lack of Efficacy | 1 | 4 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- DFMO and Etoposide: DFMO: Escalating doses of DFMO in a 3 +3 cohort design.
  DFMO at current cohort Dose Level orally each day for 21 day cycles
  Dose level 1: 500 mg/m2 PO BID Dose level 2: 750 mg/m2 PO BID Dose level 3:1000 mg/m2 PO BID Dose level 4:1500 mg/m2 PO BID
  Etoposide: Starting with Cycle 2, etoposide will be given at 50mg/m2/dose PO daily for the first 14 days of each 21 day cycle. Capsules will be rounded to closest 50 mg.
Arm/Group | DFMO and Etoposide
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 8.75 [1 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: To determine the safety, tolerability and maximum tolerated dose (MTD) of DFMO as a single agent and in combination with etoposide in pediatric and young adult patients with refractory or recurrent neuroblastoma
Time Frame: length of study plus 30 days
Population: Received at least one dose of DFMO
Measure: Number; unit: participants
Arm/Group | Dose Level 1: 500 mg/m2 PO BID | Dose Level 2: 750 mg/m2 PO BID | Dose Level 3:1000 mg/m2 PO BID | Dose Level 4:1500 mg/m2 PO BID
Number analyzed (Participants) | 4 | 5 | 3 | 9
participants | 2 | 4 | 0 | 5

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 2 years
Population: 18 subjects out of the 21 enrolled were evaluable. 3 subjects did not make it to an evaluable time point.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | DFMO and Etoposide
Number analyzed (Participants) | 18
Days | 85 [62 to 418]

3. Secondary Outcome: Number of Patients With an Overall Response Rate (ORR) of PR or CR
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Population: 18 subjects out of the 21 enrolled were evaluable. 3 subjects did not make it to an evaluable time point.
Measure: Number; unit: participants
Arm/Group | DFMO and Etoposide
Number analyzed (Participants) | 18
participants | 4

4. Secondary Outcome: Tmax of DFMO in Pediatrics Using Pharmacokinetic (PK) Testing.
Time Frame: Cycle 1 Day 8 at hour 0 (pre-dose), 30 minutes, 1 hour, 3 hours, and 6 hours
Population: Cohort at max dose of 1500mg/m2 BID
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | DFMO and Etoposide
Number analyzed (Participants) | 9
hours | 2.88 (1.45)

5. Secondary Outcome: Cmax of DFMO in Pediatrics Using Pharmacokinetic (PK) Testing.
Time Frame: Cycle 1 Day 8 at hour 0 (pre-dose), 30 minutes, 1 hour, 3 hours, and 6 hours
Population: Cohort at max dose of 1500mg/m2 BID
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | DFMO and Etoposide
Number analyzed (Participants) | 9
mcg/ml | 28.89 (14.96)

6. Secondary Outcome: AUC of DFMO in Pediatrics Using Pharmacokinetic (PK) Testing.
Time Frame: Cycle 1 Day 8 at hour 0 (pre-dose), 30 minutes, 1 hour, 3 hours, and 6 hours
Population: Cohort at max dose of 1500mg/m2 BID
Measure: Mean (Standard Deviation); unit: (mcg/ml) * hr
Arm/Group | DFMO and Etoposide
Number analyzed (Participants) | 9
(mcg/ml) * hr | 108.38 (53.23)

ADVERSE EVENTS:
Time Frame: New adverse events collected from first dose of study drug to 30 days past last dose of study drug. Related adverse events followed until resolution.
Arm/Group | DFMO and Etoposide
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 11/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFMO and Etoposide (N=21)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Back Pain unrelated to study drug.
Progression of Disease resulting in death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFMO and Etoposide (N=21)
Anemia (Blood and lymphatic system disorders) | 4 (8)
Neutorpenia (Blood and lymphatic system disorders) | 5 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (5)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
ALT elevation (Hepatobiliary disorders) | 2 (2)
Anorexia (General disorders) | 1 (1)
AST elevation (Hepatobiliary disorders) | 3 (3)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
GGT elevation (Blood and lymphatic system disorders) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 (1)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)
Infection, sinus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mouth pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep disturbance (General disorders) | 1 (1)
urinary retention (Renal and urinary disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less